CLINICAL TRIAL: NCT03152045
Title: Teaching Improved Communication To Adolescents and Clinicians
Acronym: TicTac
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Pro00078439
Record Dates: First submitted 2017-05-02; First posted 2017-05-12 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-10

CONDITIONS: Communication Improvement Between Adolescent and Clinician
Keywords: communication between adolescent patients and their clinician

STUDY DESIGN:
Intervention Model Description: Interventional: to evaluate the effect of Feedback Guides on clinician-adolescent communication about hight-risk behaviors.
  Control: standard of care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Communication Intervention (Experimental): Investigators are testing the feasibility, acceptability, and preliminary efficacy of a systems intervention that asks adolescents to report their risk behaviors before their encounter. Both clinicians and patients will receive a Feedback Guide that gives them tips on effective ways to communicate about these behaviors.
  Interventions: Behavioral: Communication Intervention
- Standard Of Care (No Intervention): Investigators will compare patients randomized into the intervention group to those who receive standard of care.

INTERVENTIONS:
Behavioral: Communication Intervention — In this study, Investigators are testing the feasibility, acceptability, and preliminary efficacy of a systems intervention that asks adolescents to report their risk behaviors before their encounter. Both clinicians and patients will receive a Feedback Guide that gives them tips on effective ways to communicate about these behaviors.
  Arms: Communication Intervention

SUMMARY:
The purpose of this pilot study is to evaluate the feasibility, acceptability, and preliminary efficacy of an intervention aimed at improving how adolescent patients and their clinicians communicate about behavior change.

DETAILED DESCRIPTION:
The investigators propose a randomized pilot trial across two health systems, Duke University and University of Michigan to evaluate the effect of Feedback Guides on clinician-adolescent communication about high-risk behaviors.

* The investigators consent clinicians prior to any patient recruitment.
* When a patient aged 12-21 years arrives for an annual visit and is a patient of a consented clinician, the front desk staff will provide the teen with an iPad tablet.
* As part of standard clinical care, all teens will complete the Rapid Assessment for Adolescent Preventive Services (RAAPS) questionnaire on the tablet privately (either in waiting room or in clinic room while waiting for the provider).
* The patient and parent will then review a study explanation and informed consent on the tablet and sign electronically if they agree to participate. The study clinician will review the informed consent with the patient and answer any questions.
* Participating teens will then complete a brief baseline survey and those randomized to the intervention arm will print the visit conversation guides using a wireless study printer connected to the tablet. The guides will print in a designated nursing area and clinic staff will add the printed guides to visit-related paperwork for the patient and clinician to use during the visit.
* The teen patient audio records the encounter on the tablet.
* The patient completes post-visit patient survey on tablet.
* The clinician completes a post-visit survey on paper.
* The patient returns tablet to clinic staff.
* The iPad will be connected to a study workstation, where the iTunes application will be used to transfer the audio file from the Voice Memos app to the workstation and then to it's final destination on the file server. Once the transfer has been confirmed, using iTunes, the audio file will be deleted from both the iPad and the workstation, including any residual versions of the audio file.
* Three months after the encounter, staff will provide participating patients a link to a REDCap survey (not the survey itself). The link will be sent using the preferred method selected by the patient through a question in the baseline survey - email or short message service (SMS). To protect the confidentiality of the responses, we will also provide the participant a code to access the REDCap follow-up survey. This will prevent others from accessing the survey results.

ELIGIBILITY:
Inclusion Criteria:

* All English-speaking adolescent patients
* cognitively able to participate

Exclusion Criteria:

* Adolescents less than 12 years of age
* Adolescents over 21 years of age
* cognitively unable to participate.

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-10-29 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by recruitment number | 9 months
  We will consider the intervention feasible if we recruit 20 adolescent patients and up to 10 clinicians per site.

SECONDARY OUTCOMES:
Acceptability | 9 months
  To determine acceptability, we will examine patients' reports of rated helpfulness of the intervention. To be deemed acceptable, 75% would have to rate it as a "4" or "5" on the 5-point scale

OTHER OUTCOMES:
Patient perceived provider empathy as measure by a summed 10-question scale | 10 minutes
  We will assess patient perceived provider empathy with a summed 10-question scale (α=0.95; e.g., "Thinking about your visit with your doctor, how was your doctor at fully understanding your concerns?" (1= Not at all good and 5= Extremely good)).
Patient perceived autonomy support using a 15 question scale | 10 minutes
  We will assess patient autonomy support using a 15 question scale (a=0.95;e.g., "I feel that my physician has provided me choices and potions" (1=Strongly disagree and 5=Strongly agree).
Patient's self rated participation in the encounter | 10 minutes
  We will assess patient's self rated participation in the encounter using a five-point Likert-type scale (i.e., 1 "Not at all good" - 5 "Extremely good")

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Pollak, PhD, Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke University Medical Center, Durham, North Carolina
  - Duke University Medical Center - Cancer Prevention, Detection and Control, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No
De-identified web-based surveys from the University of Michigan will be available to Duke researchers through REDCap.

REFERENCES:
- [Result] Hoglund AT, Winblad U, Arnetz B, Arnetz JE. Patient participation during hospitalization for myocardial infarction: perceptions among patients and personnel. Scand J Caring Sci. 2010 Sep;24(3):482-9. doi: 10.1111/j.1471-6712.2009.00738.x. PMID 20230518
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/20230518